CLINICAL TRIAL: NCT02773303
Title: Neurofeedback Therapy for Children Diagnosed With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI-IRB-20160321001
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Neurofeedback; balance, postural; postural equilibrium; EEG
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): Children receiving Mente Autism™ neurofeedback therapy to use at home for 40 minutes a day for 12 weeks
  Interventions: Device: Mente Autism™
- Control (Sham Comparator): Children not receiving neurofeedback based therapy, but receiving the Sham therapy
  Interventions: Device: Sham

INTERVENTIONS:
Device: Mente Autism™ — A portable headband records EEG activity, and specialized algorithms convert the EEG activity into sonified binaural signals feeding them back to the user
  Arms: Active
Device: Sham — a device externally identical to Mente Autism™, providing binaural beats but not tailor-made neurofeedback binaural beats
  Arms: Control

SUMMARY:
This project aims:

* to further explore the effectiveness of a novel sonified Neurofeedback management therapy for children diagnosed with Autism Spectrum Disorder (ASD)
* to determine if balance control is different before and after therapy

DETAILED DESCRIPTION:
Once the informed consent of a parent or guardian has been secured, each child will be asked to provide informed assent. If the child elects to participate in the research project, he/she is enrolled in the study and assign to one of two groups: Active Comparator or Sham Comparator. If possible, his/her ability to maintain balance is then assessed using a standard extended mCTSIB protocol (standing for 25 seconds on a hard surface/4" tall foam cushion with eyes open/closed and head neutral/turned right/left/flexed or extended) and his/her baseline qEEG are recorded. A series of questionnaires will be administered to the child and/or his/her parents/legal guardian/caretaker.

Afterward the child will be instructed to wear the prescribed device (either the Active Comparator (Mente Autism™) or the Sham Comparator (a device externally identical to Mente Autism™, providing binaural beats but not tailor-made neurofeedback binaural beats)) to use at home for 40 minutes a day for 12 weeks. At the end of the 12 weeks treatment period, the child will again be tested as at the beginning of the trial (posturography, qEEG, and questionnaires). At the end of the study, participants in the Sham Comparator group will be offered the option of receiving the full therapy.

ELIGIBILITY:
Inclusion Criteria:

* a clear diagnosis of ASD and a high starting delta wave level, as confirmed by the initial qEEG.

Furthermore, since the therapy is administered via a device requiring to be connected to a computer, tablet or phone with WiFi capabilities to work, the following are additional requirement:

* iPhone 4s or later or all iPads except first generation iPAD running OS v7 or later, or
* computer running Windows 7 or later
* Tablet running Android 4.1 or later
* Internet connection

Exclusion Criteria:

* a history of hearing impairment and co-morbidities such as Rett-Syndrome and if they get low delta wave recordings in frontal lobe with qEEG (part of the baseline testing battery)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Changes in qEEG | Baseline and at week 12
  Changes will be assessed between baseline (at enrollment) and after the treatment period. It will be used to investigate if Mente Autism™ therapy affect it and how much.

SECONDARY OUTCOMES:
Changes in Stability Score | Baseline and at week 12
  The Stability Score is calculated as percentage ratio of the actual sway and the theoretical limit of stability.
  Changes in Stability Score will be assessed between baseline (at enrollment) and after the treatment period. It will be used to investigate if Mente Autism™ therapy affect it and how much.
Changes in Questions about Behavioural Function (QABF) test | Baseline and at week 12
  Changes will be assessed between baseline (at enrollment) and after the treatment period. It will be used to investigate if Mente Autism™ therapy affect it and how much.
The Behavior Rating Inventory of Executive Function (BRIEF) | Baseline and at week 12
  Changes will be assessed between baseline (at enrollment) and after the treatment period. It will be used to investigate if Mente Autism™ therapy affect it and how much.
Changes in Social Responsiveness Scale (Second Edition) SRS-2 | Baseline and at week 12
  Changes will be assessed between baseline (at enrollment) and after the treatment period. It will be used to investigate if Mente Autism™ therapy affect it and how much.
Changes in Autism Behaviour Checklist (ABC) | Baseline and at week 12
  Changes will be assessed between baseline (at enrollment) and after the treatment period. It will be used to investigate if Mente Autism™ therapy affect it and how much.

OTHER OUTCOMES:
The Autism Treatment Evaluation Checklist (ATEC) | Baseline and at week 12
  Changes will be assessed between baseline (at enrollment) and after the treatment period. It will be used to investigate if Mente Autism™ therapy affect it and how much.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, Principal Investigator — Carrick Institute for Graduate Studies
Locations (1):
- Plasticity Brain Centers, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrick FR, Pagnacco G, Hankir A, Abdulrahman M, Zaman R, Kalambaheti ER, Barton DA, Link PE, Oggero E. The Treatment of Autism Spectrum Disorder With Auditory Neurofeedback: A Randomized Placebo Controlled Trial Using the Mente Autism Device. Front Neurol. 2018 Jul 5;9:537. doi: 10.3389/fneur.2018.00537. eCollection 2018. PMID 30026726